CLINICAL TRIAL: NCT00408330
Title: A Double-Blind, Randomized, Vehicle-Controlled, Six-Week Exploratory Multicenter Pilot Study of the Efficacy and Safety of Azelaic Acid (AzA) 15% Gel in the Topical Treatment of Mild to Moderate Seborrheic Dermatitis of the Face
Brief Title: A Study of Azelaic Acid (AzA) 15% Gel in the Treatment of Seborrheic Dermatitis of the Face
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1401201; 2006-002060-26 (EudraCT Number)
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2015-03

CONDITIONS: Seborrheic Dermatitis on the Face
MeSH Terms: interventions — azelaic acid; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): azelaic acid 15%
  Interventions: Drug: Azelaic Acid 15% Gel
- 2 (Placebo Comparator): Inactive 15% gel base
  Interventions: Drug: Inactive 15% gel base

INTERVENTIONS:
Drug: Azelaic Acid 15% Gel — 15% gel, topically applied daily for six weeks
  Arms: 1
Drug: Inactive 15% gel base — placebo, topically applied daily for six weeks
  Arms: 2

SUMMARY:
This study is to determine whether a medication on the market for other indications is effective and safe in treating seborrheic dermatitis of the face.

DETAILED DESCRIPTION:
To test the efficacy and safety of azelaic acid 15% gel in the treatment of seborrheic dermatitis of the face

ELIGIBILITY:
Inclusion Criteria:

- Stable or exacerbating seborrheic dermatitis in the facial area

Exclusion Criteria:

* Psoriasis
* Atopic dermatitis
* Facial acne and rosacea
* Dermatophytic skin infections
* Parkinson's disease
* Known immunosuppression; HIV infection
* Any condition requiring continuous systemic or topical corticosteroid or antimycotic therapy
* Continuous asthma inhalation treatment requiring > 800 mg corticosteroids
* Any severe disease likely to interfere with the conduct or the planned termination of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Sum Score of the symptoms of seborrheic dermatitis and the investigator's global assessment. | Measurement of parameters during the course of treatment (six weeks)

SECONDARY OUTCOMES:
Investigators' and patients' subjective assessment of improvement; frequency and intensity of single symptoms | Measurement of parameters during the course of treatment (six weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Germany (3):
  - Blankenfelde-Mahlow
  - Buchholz
  - Hamburg